CLINICAL TRIAL: NCT04843813
Title: Lutein and Multiple Sclerosis Experimental Study (LuMES)
Brief Title: Effects of Lutein Supplementation on Cognition and MPOD in Multiple Sclerosis Patients-
Acronym: LuMES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Division of Nutritional Sciences, University of Illinois at Urbana-Champaign (Unknown); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Naiman Khan, Assistant Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2001-2
Record Dates: First submitted 2021-04-07; First posted 2021-04-14 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Cognitive Function; Lutein
MeSH Terms: conditions — Multiple Sclerosis | interventions — Lutein

STUDY DESIGN:
Intervention Model Description: A 2-group parallel design will be employed to collect feasibility data on daily lutein supplementation over 4 months.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lutein (Experimental)
  Interventions: Dietary Supplement: Lutein
- Safflower Oil (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lutein — Participants will consume daily soft gels containing the lutein supplement.
  Arms: Lutein
Dietary Supplement: Placebo — Participants will consume daily soft gels containing the safflower oil.
  Arms: Safflower Oil

SUMMARY:
The central hypothesis is that lutein supplementation will improve MPOD and cognition. Accordingly, the specific aims are to 1) to determine the process feasibility associated with participating in 4-month lutein supplementation trial; and 2) to investigate the scientific feasibility of 4-month daily lutein supplementation on biological markers of lutein status and cognitive function among persons with MS.

DETAILED DESCRIPTION:
A two-group parallel design will be employed whereby participants will be randomly assigned to one of 2 groups. The supplementation doses 20mg/d (Group 1), and placebo (Group 2) will be consumed daily by the participant for a 4-month period. Pre-test and follow-up measures of lutein status and cognitive function will be assessed at baseline and at 4-month follow-up via laboratory visits.

ELIGIBILITY:
Inclusion Criteria:

* 18-64.9 years
* Self-reported relapsing-remitting MS (RRMS) diagnosis
* Expanded Disability Status Scale (EDSS) score between 0-3.5
* Macular Pigment Optical Density at baseline (MPOD ≤0.35)
* Score ≤55 during the Symbol Digit Modalities Test (SDMT)
* 20/20 or corrected vision
* No presence of color blindness
* No history of age-related macular degeneration
* No history of epileptic seizures

Exclusion Criteria:

* Under 18 years or over 64.9 years
* MS diagnosis other than RRMS
* Pregnancy
* Uncorrected vision
* Presence of color blindness
* PDDS score of 7 or more
* Prior diagnosis of age-related macular degeneration
* History of epileptic seizures

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-26 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Macular Pigment Optical Density | 4 months (baseline vs. follow-up)
  Changes in Macular Pigment Optical Density (log units) between groups using a macular densitometer
Attentional Accuracy | 4 months (baseline vs. follow-up)
  Changes in accuracy (%) between groups using a computerized flanker task
Attentional Reaction Time | 4 months (baseline vs. follow-up)
  Changes in reaction time (ms) between groups using a computerized flanker task
Attentional Resource Allocation | 4 months (baseline vs. follow-up)
  Changes in P3 event related potential amplitude (microvolts) between groups using a computerized flanker task
Attentional Processing Speed | 4 months (baseline vs. follow-up)
  Changes in P3 event related potential latency (ms) between groups using a computerized flanker task

CONTACTS AND LOCATIONS:
Overall Officials: Naiman Khan, PhD, Principal Investigator — University of Illinois Urbana Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martell SG, Kim J, Cannavale CN, Mehta TD, Erdman JW Jr, Adamson B, Motl RW, Khan NA. Randomized, Placebo-Controlled, Single-Blind Study of Lutein Supplementation on Carotenoid Status and Cognition in Persons with Multiple Sclerosis. J Nutr. 2023 Aug;153(8):2298-2311. doi: 10.1016/j.tjnut.2023.06.027. Epub 2023 Jun 25. PMID 37364683